CLINICAL TRIAL: NCT02850263
Title: An Observational Study to Assess the Effectiveness of Intravitreal Aflibercept in Routine Clinical Practice tn Patients With Visual Impairment Due to Diabetic Macular Oedema (DMO)
Brief Title: A Study to Assess the Effectiveness of Aflibercept in Routine Clinical Practice in Patients With Diabetic Macular Oedema
Acronym: DRAKO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18058
Record Dates: First submitted 2016-05-19; First posted 2016-07-29 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Macular Edema
Keywords: Diabetic Retinopathy; Diabetic Macular Oedema; Diabetic Macular Edema; Aflibercept
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 / Anti-VEGF treatment naïve patients: Anti-VEGF treatment of naïve patients (who have not received any previous anti-VEGF treatment) with visual impairment due to diabetic macular oedema (DMO) in routine clinical practice in the United Kingdom.
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)
- Cohort 2 / Anti-VEGF treatment non-naïve patients: Anti-VEGF treatment of non-naïve patients (who have received previous anti-VEGF treatment) with visual impairment due to diabetic macular oedema (DMO) in routine clinical practice in the UK.
  Interventions: Drug: Anti-VEGF therapies including: Eylea Aflibercept, VEGF Trap-Eye, BAY86-5321) and Ophthalmologicals / Antineovascularisation agents (S01LA05)
- Cohort 3 / Total study population: Anti-VEGF treatment naïve patients and anti-VEGF treatment non-naïve patients with visual impairment due to diabetic macular oedema (DMO) in routine clinical practice in the UK.
  Interventions: Drug: Anti-VEGF therapies including: Eylea Aflibercept, VEGF Trap-Eye, BAY86-5321) and Ophthalmologicals / Antineovascularisation agents (S01LA05)

INTERVENTIONS:
Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321) — Anti-VEGF exposure is defined as treatment with intravitreal aflibercept for the treatment of DMO by the patient.according to the prescribing physician.
  Groups: Cohort 1 / Anti-VEGF treatment naïve patients
Drug: Anti-VEGF therapies including: Eylea Aflibercept, VEGF Trap-Eye, BAY86-5321) and Ophthalmologicals / Antineovascularisation agents (S01LA05) — Anti-VEGF exposure is defined as treatment with intravitreal aflibercept or another agent [Ophthalmologicals / Antineovascularisation agents (S01LA05)] for the treatment of DMO by the patient.according to the prescribing physician.
  Groups: Cohort 2 / Anti-VEGF treatment non-naïve patients
Drug: Anti-VEGF therapies including: Eylea Aflibercept, VEGF Trap-Eye, BAY86-5321) and Ophthalmologicals / Antineovascularisation agents (S01LA05) — Anti-VEGF exposure is defined as treatment with intravitreal aflibercept or another agent [Ophthalmologicals / Antineovascularisation agents (S01LA05)] for the treatment of DMO by the patient.according to the prescribing physician.
  Groups: Cohort 3 / Total study population

SUMMARY:
Intravitreal aflibercept has been approved for the treatment of visual impairments due to diabetic macular oedema (DMO) in Europe and the US in August 2014 and July 2014 respectively.

The main objectives of this observational cohort field study are to evaluate effectiveness of intravitreal aflibercept and to describe follow-up as well as treatment patterns in anti vascular endothelial growth factor (anti-VEGF) treatment naïve patients with DMO in routine clinical practice in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients diagnosed with type 1 or 2 diabetes mellitus.
* Patients diagnosed with DMO with central involvement (defined as the area of the centre subfield of OCT) treated with intravitreal aflibercept (in accordance with routine practice).
* Patients for whom the decision to initiate treatment with intravitreal aflibercept was made as per the investigator's routine treatment practice and prior to study inclusion.
* Patients must provide written informed consent.

Exclusion Criteria:

* Patients under the age of 18.
* Patients with contraindications as listed in the SmPC for intravitreal aflibercept.
* Patients with pre-planned cataract surgery during the observational period.
* Patients previously treated with intravitreal anti-VEGF within 28 days.
* Patients currently or previously treated with systemic anti-VEGF.
* Patients previously treated with intravitreal fluocinolone acetonide steroid.
* Patients participating in an investigational programme with interventions outside of routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients with a diagnosis of diabetic macular oedema with central involvement will be enrolled after the decision for treatment with intravitreal aflibercept has been made.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) in Early Treatment Diabetic Retinopathy Study (ETDRS) letters in patients with DMO treated with intravitreal aflibercept | Baseline and 12 months
  BCVA (Best Corrected Visual Acuity): process to measure with the help of a retinoscope, auto-refractor or phoropter how much power is needed to bring the eye to normal, perfectly focused vision) when performed in addition to that at baseline and 12 months. ETDRS Chart: charts imprinted with lines of letters decreasing in size from largest on top to smallest on the bottom to determine visual acuity.
Change in central subfield thickness (CST) as determined by Spectral Domain Optical Coherence Tomography (SD-OCT) in patients with DMO treated with intravitreal aflibercept | Baseline and 12 months

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) in Early Treatment Diabetic Retinopathy Study (ETDRS) letters in patients with DMO treated with intravitreal aflibercept | Baseline and 24 months
Change in central subfield thickness (CST) as determined by Spectral Domain Optical Coherence Tomography (SD-OCT) in patients with DMO treated with intravitreal aflibercept | Baseline and 24 months
Change in non-refracted visual acuity in patients with DMO treated with intravitreal aflibercept | Baseline, 12 and 24 months
Change in Best Corrected Visual Acuity (BCVA) in Early Treatment Diabetic Retinopathy Study (ETDRS) letters in patients with DMO treated with intravitreal aflibercept differentiated by BCVA baseline characteristics | Baseline, 12 and 24 months
Change in central subfield thickness (CST) in patients with DMO treated with intravitreal aflibercept differentiated by CST baseline characteristics | Baseline, 12 and 24 months
Proportion (%) of patients discontinuing intravitreal aflibercept treatment | Baseline, 12 and 24 months
Time between the decision to treat for patients with DMO who have not received any previous anti-VEGF treatment | Baseline
The time between the date of DMO diagnosis for patients with DMO who have received any previous anti-VEGF treatment | Baseline
Proportion (%) of treated eyes with 5, 10 and 15 letter gain / loss | Baseline, 12 and 24 months
Proportion (%) of sites that adhere to their stated treatment protocol | 12 and 24 months
Change in QoL score measured by NEI VFQ-25 | Baseline, 12 and 24 months
Change in macular volume | Baseline, 12 and 24 months
Change in Best Corrected Visual Acuity (BCVA) in Early Treatment Diabetic Retinopathy Study (ETDRS) letters | Baseline, 12 and 24 months
Change in non-refracted visual acuity (VA).for the fellow eye | Baseline, 12 and 24 months
Number of DMO treatments required for the fellow eye | Baseline, 12 and 24 months
Number of visits performed (resources) to assess the fellow eye | Baseline, 12 and 24 months
Number of clinical procedures performed (resources) to assess the fellow eye | Baseline, 12 and 24 months
Number of adverse events as a measure of safety and tolerability | 24 months
Reason for discontinuation of intravitreal aflibercept treatment | Baseline, 12 and 24 months
Change in Central Subfield Thickness (CST) of the fellow eye | Baseline, 12 and 24 months
Type of DMO treatments required for the fellow eye | Baseline, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Sivaprasad S, Ghanchi F, Kelly SP, Kotagiri A, Talks J, Scanlon P, McGoey H, Nolan A, Saddiq M, Napier J; DRAKO study group. Evaluation of standard of care intravitreal aflibercept treatment of diabetic macular oedema treatment-naive patients in the UK: DRAKO study 12-month outcomes. Eye (Lond). 2022 Jan;36(1):64-71. doi: 10.1038/s41433-021-01624-9. Epub 2021 Jul 9. PMID 34244670
- [Derived] Sivaprasad S, Ghanchi F, Kelly SP, Kotagiri A, Talks J, Scanlon P, McGoey H, Nolan A, Saddiq M, Napier J. Evaluation of care with intravitreal aflibercept treatment for UK patients with diabetic macular oedema: DRAKO study 24-month real-world outcomes. Eye (Lond). 2023 Sep;37(13):2753-2760. doi: 10.1038/s41433-023-02409-y. Epub 2023 Mar 20. PMID 36941402